CLINICAL TRIAL: NCT01080248
Title: A Phase II Study of Gemcitabine and Pazopanib in Metastatic Pancreatic Cancer
Brief Title: Gemcitabine and Pazopanib in Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to delay by GSK
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-0434 / 201103201
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-05

CONDITIONS: Pancreatic Cancer
Keywords: Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (gemcitabine & pazopanib) (Experimental): Gemcitabine 1000 mg/m2 IV on days 1, 8, and 15 of each 28 day cycle.
  Pazopanib 800 mg PO daily of each 28 day cycle.
  Interventions: Drug: Gemcitabine; Drug: Pazopanib

INTERVENTIONS:
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Pazopanib
  Other Names: Votrient

SUMMARY:
To determine the response rate and survival of gemcitabine and pazopanib in patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
To determine the response rate by RECIST criteria.

To determine the progression free survival.

To determine the median survival and overall survival at one year.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma.
* Patient must have metastatic disease that is not amenable to surgical resection.
* Patient must have measurable disease (by RECIST criteria), defined as at least one lesion that can be accurately measured in at least one dimension.
* Patient may have previously untreated disease or may have been previously treated if they meet the following criteria:

  * received adjuvant gemcitabine therapy >6 months prior to enrollment with progression off therapy
  * received prior radiation therapy > 4 weeks prior to study enrollment and have measurable tumor mass outside the radiation field
  * received prior radiation therapy > 4 weeks prior to study enrollment, have a measurable tumor mass outside the radiation field, and received 5-FU as a radiation sensitizer >4 weeks prior to study enrollment
* Patient must be >=18 years old. Note: pazopanib is contraindicated in the pediatric population due to the potential effect on the epiphyseal growth plates.
* Patient must have an ECOG performance status of 0-1
* Patient must have normal organ and marrow function within 14 days of study initiation as defined below:

  * ANC ≥ 1.5 x 109/L
  * Hemoglobin ≥ 9 g/dL; patients may not have had a transfusion within 7 days of screening assessment
  * Platelets ≥ 100 x 109/L
  * PT or INR ≤ 1.2 x upper limit of normal (ULN)
  * PTT ≤ 1.2 x ULN
  * Total bilirubin ≤ 1.5 x ULN
  * AST and ALT ≤ 2.5 x ULN
  * Serum creatinine ≤ 1.5 mg/dL; if > 1.5 mg/dL, calculated creatinine clearance must be ≥ 50 mL/min
  * Urine protein to creatinine ratio < 1; if ≥ 1, then a 24-hour urine protein must be assessed and must be < 1 g in order for patients to be eligible
* Patient must have the ability to understand and the willingness to sign a written informed consent document.
* Eligible patients of reproductive potential (both sexes) must agree to use adequate contraceptive methods.

Exclusion Criteria

* Patient has been treated with an agent that antagonizes the VEGF receptor.
* Patient has received any other investigational agents < 28 days prior to enrollment.
* Patient has known brain metastases; these patients are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. In addition, patients with brain metastases may be at a higher theoretical risk for cerebral hemorrhage while taking pazopanib.
* Patient has a history of allergic reactions attributed to compounds of similar chemical or biologic composition to pazopanib, gemcitabine, or other agents used in the study.
* Patient has an increased risk of hemorrhage such as having received thrombolytic agents within the past month, being on an unstable dose of anticoagulation, or having a known bleeding diathesis.
* Patient has a clinically significant gastrointestinal abnormality that may increase the risk for GI bleeding such as:

  * Active inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease) or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess ≤ 28 days prior to beginning study treatment
* Patient has a history of any one or more of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Coronary artery by-pass graft surgery
  * Symptomatic peripheral vascular disease
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Patient has prolonged QT intervals, taking antiarrhythmics or taking other medications that prolong QT
* Patient has poorly controlled hypertension (defined as systolic blood pressure (SBP) of ≥160 mmHg or diastolic blood pressure (DBP) of ≥ 90 mmHg). Note: initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry.
* Patient has a history of cerebrovascular accident, pulmonary embolism, or untreated deep venous thrombosis (DVT) within the past 6 months.
* Patient has had major surgery, trauma, non-healing wound, fracture, or ulcer within 28 days prior to first dose of gemcitabine and/or study drug (procedures such as catheter placement not considered to be major) OR minor surgery within 14 days prior to first dose of gemcitabine and/or study drug.
* Patient has significant proteinuria as evidenced by urine protein/creatinine ratio >1
* Patient has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, cardiac arrhythmia, active second malignancy, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patient is pregnant or breastfeeding. Pregnant women are excluded from this study because pre-clinical reproductive toxicity studies with pazopanib demonstrated reduced female fertility and teratogenic effects.
* Patient is known HIV-positive. These patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Patient is a known alcohol, cocaine, or IV drug abuser within 6 months prior to enrollment.
* Patient is receiving treatment with any of the following anti-cancer therapies:

  * Radiation therapy, surgery, or tumor embolization within 4 weeks prior to the first dose of pazopanib OR
  * Chemotherapy, immunotherapy, biologic therapy, investigational therapy, or hormonal therapy within 28 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib.
* Patient is experiencing any ongoing toxicity from prior anti-cancer therapy that is > grade 1 and/or that is progressing in severity.
* Inclusion of Women and Minorities
* Both men and women and members of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Picus, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 08/26/2010 and closed to participant enrollment on 09/27/2011.
Period: Overall Study
Arm/Group | Arm 1 (Gemcitabine & Pazopanib)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1 (Gemcitabine & Pazopanib)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Response Rate by RECIST Criteria.
Description: * Response rate = complete response + partial response per RECIST
  * Complete response - disappearance of all target and non-target lesions.
  * Partial response - at least a 30% decrease in the sum of the longest diameter of the target lesions, taking as reference the baseline sum longest diameter
Time Frame: Follow-up was approximately 9 weeks
Population: One participant was removed from study for adverse event prior to first response assessment. The remaining participant had progressive disease per RECIST while on treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 (Gemcitabine & Pazopanib)
Number analyzed (Participants) | 1
percentage of participants | 0

2. Secondary Outcome: Progression-free Survival (PFS)
Description: * PFS is defined as the duration of time from start of treatment to time to progression.
  * Progressive disease - at least a 20% increase in the sum of the longest diameter of the target lesions taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Follow-up was approximately 9 weeks
Population: One participant was removed from study for adverse event prior to first response assessment.
Measure: Number; unit: weeks
Arm/Group | Arm 1 (Gemcitabine & Pazopanib)
Number analyzed (Participants) | 1
weeks | 8

3. Secondary Outcome: Median Survival
Time Frame: Length of follow-up was 35 weeks
Measure: Median (Full Range); unit: weeks
Arm/Group | Arm 1 (Gemcitabine & Pazopanib)
Number analyzed (Participants) | 2
weeks | 34 [33 to 35]

4. Secondary Outcome: Overall Survival
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Arm 1 (Gemcitabine & Pazopanib)
Number analyzed (Participants) | 2
participants | 0

ADVERSE EVENTS:
Arm/Group | Arm 1 (Gemcitabine & Pazopanib)
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (Gemcitabine & Pazopanib) (N=2)
Alkaline phosphatase (Investigations) | 1
Bloating (Gastrointestinal disorders) | 1
Chills (General disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema (General disorders) | 1
Fatigue (General disorders) | 2
Fever (General disorders) | 1
Gastrointestinal bleed (Gastrointestinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 1
Pain (General disorders) | 1
SGOT/SGPT (Investigations) | 2
Sweating (General disorders) | 2
Urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
Granulocytes (Investigations) | 1
Hemoglobin (Blood and lymphatic system disorders) | 2
Leukopenia (Investigations) | 2
Platelets (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes